CLINICAL TRIAL: NCT00646659
Title: Randomized Phase II Feasibility Study of Cetuximab Combined With 4 Cycles of TPF Followed by Platinum Based Chemo-radiation Strategies
Brief Title: Cetuximab, Combination Chemotherapy, and Radiation Therapy in Treating Patients With Newly Diagnosed Stage III or Stage IV Head and Neck Cancer That Cannot Be Removed By Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment was suspended prematurely for safety concerns and closed after IDMC review
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-24061; MERCK-EORTC-24061; SANOFI-AVENTIS-EORTC-24061; 2006-004189-14 (EudraCT Number)
Record Dates: First submitted 2008-03-27; First posted 2008-03-28 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; untreated metastatic squamous neck cancer with occult primary
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Carboplatin; Cisplatin; Docetaxel; Fluorouracil; In Situ Hybridization, Fluorescence; Genetic Testing; Reverse Transcriptase Polymerase Chain Reaction; Immunoenzyme Techniques; Immunohistochemistry; Biopsy; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

INTERVENTIONS:
Biological: cetuximab
Drug: carboplatin
Drug: cisplatin
Drug: docetaxel
Drug: fluorouracil
Genetic: fluorescence in situ hybridization
Genetic: molecular genetic technique
Genetic: reverse transcriptase-polymerase chain reaction
Other: immunoenzyme technique
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: biopsy
Radiation: 3-dimensional conformal radiation therapy
Radiation: intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may also stop the growth of tumor cells by blocking blood flow to the tumor. Radiation therapy uses high energy x- rays to kill tumor cells. Cetuximab may also make tumor cells more sensitive to radiation therapy. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known which regimen of radiation therapy, combination chemotherapy, and cetuximab and is most effective in treating patients with head and neck cancer.

PURPOSE: This randomized phase II trial is comparing two different regimens of radiation therapy given together with combination chemotherapy and cetuximab to see how well they work in treating patients with newly diagnosed stage III or stage IV head and neck cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the safety profile of chemoradiotherapy with carboplatin vs cisplatin in patients with newly diagnosed, unresectable stage III or IV squamous cell carcinoma of the head and neck.
* To select one of these chemoradiotherapy regimens to be used as an experimental arm in a future phase III trial.
* To look for EGFR expression and downstream signaling in reacting skin samples from patients experiencing skin toxicity and in normal skin samples from the same patients for comparison with skin samples from patients who have not shown skin toxicity.
* To explore which factors related to EGFR predict the biological activity of cetuximab in patients treated with these regimens.

OUTLINE: This is a multicenter study.

Patients receive induction chemotherapy comprising docetaxel IV over 1 hour and cisplatin IV over 1 hour on day 1 and fluorouracil IV continuously over 24 hours on days 1-5. Treatment repeats every 3 weeks for up to 4 courses in the absence of unacceptable toxicity.

Within 3 weeks after completion of induction chemotherapy or within 5 weeks from the start of the last chemotherapy course (day 21), patients are stratified by institution and treatment response (stable disease [SD], partial response [PR], or complete response [CR] vs non-response [progressive disease]). Patients with progressive disease are removed from study and patients with SD, PR, or CR are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo radiotherapy (RT) (3-dimensional conformal RT or intensity-modulated RT) on days 1-5 weekly for up to 7 weeks. Beginning on day 1 of RT, patients receive cisplatin IV over 1 hour once weekly for up to 7 weeks.
* Arm II: Patients undergo RT as in arm I. Beginning on day 1 of RT, patients receive carboplatin IV over 1 hour once weekly for up to 7 weeks.

Patients in both arms receive cetuximab IV over 1-2 hours once weekly beginning on day 1 of induction chemotherapy and continuing until the end of concurrent chemoradiotherapy.

Primary tumor tissue and skin biopsies, including fixed paraffin-embedded tissue specimens or frozen tissue, are collected at baseline (prior to treatment) and after completion of study treatment for correlative laboratory studies of EGFR expression and downstream signaling. Specimens are assessed by immunohistochemistry, fluorescence in situ hybridization, and reverse transcriptase-PCR sequencing of genes and proteins for ErbB-related activation. In the event of skin toxicity during treatment, patients undergo at least two additional biopsies, one in reacting skin and one in normal skin. Samples are assessed for markers of treatment efficacy related to cetuximab.

After completion of study therapy, patients are followed at 3 months and periodically thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed squamous cell carcinoma of the head and neck

  * Stage III or IV disease
  * Unresectable disease
* Unidimensionally or bidimensionally measurable disease
* Skin and tumor material must be available for EGFR status and downstream signaling studies
* No nasopharyngeal, nasal, or paranasal cancer
* No distant metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times the upper limit of normal (ULN)
* Alkaline phosphatase and transaminases ≤ 2.5 times ULN
* Serum creatinine ≤ 120 μmol/L (1.36 mg/dL)
* Creatinine clearance ≥ 60 mL/min
* Normal cardiac function (i.e., LVEF ≥ 50%)
* Clinically satisfactory 12-lead ECG
* No serious cardiac illness or medical condition within the past 6 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No current malignancies at other sites with the exception of cone-biopsied carcinoma of the cervix and adequately treated basal or squamous cell skin carcinoma or other cancer from which the patient has been disease-free for at least the past five years
* No unstable systemic diseases
* No active uncontrolled infections
* No psychological, familial, sociological, or geographical condition that would preclude compliance with the study protocol and follow-up schedule

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior treatment for head and neck cancer
* No other concurrent anticancer therapy
* No other concurrent investigational agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-02; Primary Completion 2010-05 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of the chemoradiotherapy part of the treatment, assessed as at least 80% dose intensity of any of the radiotherapy, the platinum, and cetuximab during the chemoradiotherapy part of the treatment

SECONDARY OUTCOMES:
Toxicity as assessed by NCI CTCAE v3.0
Dose modifications
Response rate (complete or partial response)
EGFR expression and downstream signaling in primary tumor and in skin samples

CONTACTS AND LOCATIONS:
Overall Officials: Jan B. Vermorken, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium